CLINICAL TRIAL: NCT07145892
Title: Three-dimensional Digital Breast Tomosynthesis Versus Digital Mammography: Which Get the Supremacy in Diagnosis of Benign Breast Lesions in Asymptomatic Females
Brief Title: Three-dimensional Digital Breast Tomosynthesis Versus Digital Mammography
Status: Completed | Type: Observational
Sponsor: The General Authority for Teaching Hospitals and Institutes (Network)
Responsible Party: Principal Investigator, Hekmat Samir Baumey, Lecturer of Diagnostic Radiology, Damnhour National Medical Institute, The General Authority for Teaching Hospitals and Institutes
Other Study IDs: HD000217
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Three Dimension; Digital Tomosynthesis; Digital Mammography; Diagnosis; Benign Breast Lesions; Asymptomatic Females
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I: Categorized 130 women aged from 30 to 40 years.
  Interventions: Device: Three-dimensional Digital Breast Tomosynthesis; Device: Two-dimensional Digital Mammography
- Group II: Categorized 115 women aged from 40 to 50 years.
  Interventions: Device: Three-dimensional Digital Breast Tomosynthesis; Device: Two-dimensional Digital Mammography
- Group III: Categorized 10 females aged above 50 years.
  Interventions: Device: Three-dimensional Digital Breast Tomosynthesis; Device: Two-dimensional Digital Mammography

INTERVENTIONS:
Device: Three-dimensional Digital Breast Tomosynthesis — Patients underwent three-dimensional digital breast tomosynthesis.
Device: Two-dimensional Digital Mammography — Patients underwent two-dimensional digital mammography

SUMMARY:
This study aimed to compare the supremacy of (3D) tomosynthesis versus (2D) digital mammography in the diagnosis of benign breast lesions in asymptomatic females.

DETAILED DESCRIPTION:
Most of the breast lesions are benign, but much concern is given to malignant lesions because breast cancer is the most common malignancy in women.

Mammography is the only study for screening in asymptomatic patients, and it is the initial imaging study in the diagnosis of symptomatic patients, with a sensitivity for suspicious lesions of 86% and a specificity of 57%.

In recent years, a significant effort has been expended to develop new approaches to breast imaging, one of which is the use of digital breast tomosynthesis (DBT), which is a pseudo three-dimensional digital mammography system that produces a series of thin-section reconstructed images from low-dose X-ray projections at multiple angles.

ELIGIBILITY:
Inclusion Criteria:

- Women with benign breast lesions.

Exclusion Criteria:

* Pregnant and lactating female.
* Patients who refuse to fill the consent form.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with benign breast lesions
Study Population: This retrospective study was conducted on patients referred to the Diagnostic Radiology Department at Damanhur Educational Hospital and Tanta University.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Correlation between imaging findings and the final diagnosis | 6 months post-procedure
  Correlation between imaging findings and the final diagnosis was calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- General Authority for Teaching Hospitals and Institutes, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.